CLINICAL TRIAL: NCT00254592
Title: Neoadjuvant Biweekly Doxorubicin and Cyclophosphamide With GMCSF Followed by Weekly Carboplatin/Nab-paclitaxel Plus or Minus Trastuzumab and Plus or Minus Bevacizumab in Treatment of Large or Inflammatory Breast Cancer-a Phase II Study
Brief Title: Neoadjuvant Treatment of Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Rita Sanghvi, Mehta, Clinical Professor, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCI 05-38; 2005-4550 (Other: University of California, Irvine)
Record Dates: First submitted 2005-11-15; First posted 2005-11-16 (Estimated); Results first posted 2013-11-11 (Estimated); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Breast Cancer
Keywords: Inflammatory; Breast Cancer; Female; Neo-adjuvant; HER-2 positive; Hormone receptor
MeSH Terms: conditions — Breast Neoplasms | interventions — Doxorubicin; Cyclophosphamide; Carboplatin; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim; Trastuzumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- AC with GM-CSF and Carboplatin/Nab-Paclitaxel (Experimental): Doxorubicin and cyclophosphamide (AC) administered intravenously every 14 days up to a total of 4 cycles, with GM-CSF on days 4-13, depending on tumor response.
  Two weeks after the completion of AC, weekly doses of carboplatin/nab-paclitaxel will be given for 3 weeks, followed by 1 week of rest, for a total of 9-12 doses. Subjects who receive 4 cycles of AC will receive 9 doses of nab-paclitaxel and subjects who receive 2 cycles of AC will receive 12 weeks of nab-paclitaxel. In addition, subjects will receive trastuzumab weekly (12-16) doses if they are Her-2 positive and bevacizumab (6-8) doses every 2 weeks if they are Her-2 negative. Each clinic visit will last approximately ½ hour.
  Interventions: Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Carboplatin; Drug: Nab-paclitaxel; Drug: GM-CSF; Drug: Trastuzumab; Drug: Bevacizumab

INTERVENTIONS:
Drug: Doxorubicin — 60 mg/m2 IV, bolus once a day every 14 days x 2-4 cycles
  Other Names: Adriamycin; NSC-123127
Drug: Cyclophosphamide — 600 mg/m2 IV once a day every 14 days x 2-4 cycles
  Other Names: Cytoxan; NSC-26271
Drug: Carboplatin — AUC 2 IV weekly for 9-12 doses beginning two weeks after completion of last AC dose
  Other Names: Paraplatin; NSC 241240
Drug: Nab-paclitaxel — 100 mg/m2 IV over 30 min weekly for 9-12 doses beginning two weeks after completion of last AC dose
  Other Names: Albumin-stabilized nanoparticle formulation of paclitaxel; Abraxane; ABI 007
Drug: GM-CSF — 250 μg/mL IV or on day 4-13 of each subcutaneous cycle of doxorubicin and injection cyclophosphamide
  Other Names: Sargramostim; Leukine; Berlex; NSC-613795
Drug: Trastuzumab — 4mg/kg, and then2 mg/kg q wk IV weekly for 12-16 doses beginning two weeks after completion of last AC dose
Drug: Bevacizumab — 10mg/kg q 2 wks
  Other Names: Avastin

SUMMARY:
Study Aims

1. To measure the clinic response rates in patients with breast cancer more than 2 cm and/or lymph node positive breast cancer treated with 2-4 cycles of biweekly doxorubicin, cyclophosphamide with Granulocyte-macrophage colony-stimulating factor (GM-CSF) (days 4-13) followed by weekly carboplatin/nab-paclitaxel given for 3 weeks, followed by 1 week of rest, for a total of 9-12 doses. (Her-2 positive patients, in addition, will receive Trastuzumab weekly (12-16 doses) and Her-2 negative patients will receive Bevacizumab (6-8 doses) q 2 weeks).
2. To measure the microscopic pathological response rate of this regimen.
3. To measure toxicity and the delivered dose intensity of this regimen.
4. To assess the association between microscopic pathologic complete response and clinical complete response at the primary tumor site in these patients.
5. To determine whether the GM-CSF increases the post treatment dendritic cells (S100+) percentage in the tumor draining lymph node as compared to pretreatment S100+ cells.
6. To determine whether the patients with a higher percent S100+ have a better clinical, pathological response, Disease Free Survival (DFS), and overall Survival (OS).
7. To determine whether flow cytometry of dendritic cells performed post-treatment in blood sample shows an increase in dendritic cell population compared to pretreatment levels.

DETAILED DESCRIPTION:
Background

Neoadjuvant chemotherapy, also termed primary, induction, or preoperative chemotherapy, is defined as chemotherapy administered before locoregional treatment. It was first used in locally advanced breast cancer 30 years ago. Classically, these tumors were treated with radical surgery and/or radiotherapy. However, despite this aggressive local therapy, most patients relapsed with distant metastases and eventually died. The aim of neoadjuvant therapy is to reduce the tumor volume in patients before surgical resection, thus increasing the likelihood of breast conservation. More recently, neoadjuvant therapy has been studied as a way of testing the relevance of biological markers in predicting disease outcome.

At least six randomized trials have compared survival in patients managed with either the neoadjuvant or adjuvant approaches. Two of the smaller trials suggested a survival advantage for patients treated with neoadjuvant chemotherapy. Other studies, including the largest trial (1,523 patients) run by the National Surgical Adjuvant Breast and Bowel Project (NSABP), found no differences in disease-free and overall survival.

Induction of a Polymerase chain reaction (pCR) should be one of the primary goals of neoadjuvant therapy because patients with no evidence of tumor cells in breast and lymph nodes after treatment may have a longer disease-free and overall survival.

Biweekly and weekly regimens may enhance dose intensity by minimizing re-growth of cells between cycles of treatment. In fact, dose dense regimens have even shown a survival benefit in an adjuvant setting in lymph node positive breast cancer, made possible with the use of G-CSF. There is no best standard neoadjuvant treatment yet. Generally patients receive AC (NSABP 14) on 3-weekly regimens in the neoadjuvant setting. In addition, incorporation of taxanes on a 3 weekly schedule has resulted in statistically higher pathological CR. More recently, weekly paclitaxel regimens have reported increased pathological responses compared to 3 weekly taxane regimens. Carboplatin has also emerged as an effective agent in the treatment of metastatic breast cancer. Moreover, the combination of carboplatin and paclitaxel has been found to be synergistic both in three-weekly regimens and weekly regimens. In fact, the combination of carboplatin, paclitaxel and trastuzumab has demonstrated a survival advantage over paclitaxel and trastuzumab alone. The Phase III study, which the preliminary results were presented at the San Antonio Breast Cancer Symposium, show that the addition of carboplatin to trastuzumab and paclitaxel resulted in a six-month improvement in the time it took for the disease to progress, compared to the standard trastuzumab and paclitaxel regimen. The study found the median survival in the trastuzumab and paclitaxel arm was 33.5 months, while the group receiving the tripartite therapy had yet to reach that point after 36 months of follow-up. Furthermore, the weekly regimens of these drugs have been found to have significantly improved tolerability over three weekly regimens. Therefore, we propose to use 2-4 cycles of AC q 2 weeks, as used in the dose dense adjuvant study with GM-CSF support on days 4-13 of the cycle. After the completion of AC we plan to administer taxol and carboplatin weekly for a total of 9-12 doses with a one-week rest after every 3 weeks of treatment over 12 weeks.

Patients who are her-2 overexpressors by FISH will also receive trastuzumab with weekly carboplatin and paclitaxel since this combination has been found to be synergistic in advanced breast cancer with improved clinical outcome. In a small study, higher pathological response rates were achieved in patients who received trastuzumab with chemotherapy compared to chemotherapy alone in the neoadjuvant. This study had a total of 34 patients who completed therapy. One arm received neoadjuvant chemotherapy with four cycles of paclitaxel followed by four cycles of fluorouracil, epirubicin, and cyclophosphamide. In the second arm, the patients received the same chemotherapy regimen with the addition of trastuzumab on a weekly schedule for twenty-four weeks. A pCR was achieved at 65.2% in the trastuzumab plus chemotherapy compared to 25% in the chemotherapy alone arm.

In metastatic breast cancer, the administration of bevacizumab to capecitabine has shown in a significant increase in response rates. The combination arm of bevacizumab plus capecitabine demonstrated a response rate of 19.8% compared to 9.1% in the capecitabine arm alone. However, the prolonged free survival or overall survival were comparable in both treatment arms. In a separate trial, the addition of bevacizumab to standard chemotherapy regimen (carboplatin and paclitaxel) in patients with advanced or relapsed non-small cell lung cancer demonstrate improved overall response and time to progression. In the bevacizumab plus standard chemotherapy, higher response rates (31.5% vs. 18.8%), longer median time to progression (7.4 vs. 4.2 months), and a modest increase in survival (17.7 vs. 14.9 months were found).

In a press release, South San Francisco, California, and Basil, Switzerland on March 14, 2005, an interim analysis of a Phase III trial showed bevacizumab plus paclitaxel and carboplatin improved overall survival compared to chemotherapy alone as a first-line therapy for non-squamous, non-small cell lung cancer. These results were presented at the American Society of Clinical Oncology (ASCO) meeting, May 13-17, 2005. This was a randomized, controlled, multicenter trial that enrolled 878 patients who had not received previous chemotherapy for non-small cell lung cancer, and compared standard chemotherapy with paclitaxel and carboplatin with or without bevacizumab. The trial was sponsored by the National Cancer Institute (NCI), part of the National Institutes of Health, under a Cooperative Research and Development Agreement between NCI and Genentech, Inc., and conducted by the Eastern Cooperative Oncology Group (ECOG).

At the San Antonio Breast Cancer Conference on December 8, 2004, Dr. Mehta et al. presented the sequential use of doxorubicin and cyclophosphamide (AC) followed by paclitaxel, carboplatin, and trastuzumab (TCH) in patient with Her-2 positive breast cancer. A pathological complete remission (pCR) was seen in 7 of 8 patients. All patients received 2-4 cycles of AC followed by 4 cycles of 3 weekly TCH regimens. Only 1 of 8 patients had a 3mm residual invasive carcinoma in the biopsy scan. Moreover, 7 of 7 patients with palpable lymph nodes demonstrated no residual cancer after this neoadjuvant regimen.

On April 18, 2005, an interim analysis of the first Phase III randomized study confirmed a significant benefit in the use of bevacizumab as first-line treatment for metastatic breast cancer. This multi-center study enrolled 722 women with previously untreated metastatic breast cancer and randomized the patients to receive adjuvant paclitaxel with or without bevacizumab. The trial excluded women who had her-2/neu positive breast cancer unless they received trastuzumab previously or were unable to receive this medication. The interim analysis showed a progression-free survival and early indication of survival benefit with the addition of bevacizumab to chemotherapy compared to chemotherapy alone. These findings were presented at ASCO this year.

In a separate trial, GM-CSF was used in breast cancer patients treated with adriamycin based chemotherapy as the preferred growth factor in a neoadjuvant setting. The initial results are suggestive of improved survival of breast cancer patients given 6 versus 5 versus 4 cycles of chemotherapy with GM-CSF support. Higher dendritic cell (DC) trafficking showed a trend toward improved survival. Moreover, patient comparison before and after treatment showed that the percentage of S100+ DC significantly increased over the course of GM-CSF treatment. The results form the basis of current hypothesis that the primary tumor may be an in vivo antigenic stimulus for dendritic cell trafficking, and that the combination of prolonged neoadjuvant chemotherapy with GM-CSF induced immune enhancement may contribute to better tumor control and better survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be women with a histologically confirmed diagnosis of breast cancer that is more than 2 cm and/or lymph node positive. Histologic confirmation shall be by either core needle biopsy or incisional biopsy. Punch biopsy is allowed if invasive breast cancer is documented.
* Patients must meet one of the criteria defined below (indicate one):

  1. Selected Stage IIB (T3, N0, M0) or IIIA (T3, N1-2, M0) disease judged primarily unresectable by an experienced breast surgeon; or otherwise deemed - appropriate candidates for neoadjuvant treatment.
  2. Stage IIIB (T4, Any N, M0) or (Any T, N3, M0) disease.
* Physical examination, chest x-ray and any x-rays or scans needed for tumor assessment must be performed within 90 days prior to registration.
* All patients must have a multiple gated acquisition (MUGA) scan or echocardiogram scan performed within 90 days prior to registration and left ventricular ejection fraction (LVEF) percentage must be greater than the institutional lower limit of normal.
* Patients must have a serum creatinine and bilirubin ≤ the institutional upper limit of normal, and an serum glutamate oxaloacetate transaminase (SGOT) or serum glutamate pyruvate transaminase (SGPT) ≤ 2x the institutional upper limit of normal. These tests must have been performed within 90 days prior to registration.
* Patients must have an absolute neutrophil count (ANC) of ≥ 1,500/μl and a platelet count of ≥ 100,000/μl. These tests must have been performed within 90 days prior to registration.
* Patients must have a performance status of 0-2 by Zubrod criteria
* In calculating days of tests and measurements, the day a test or measurement is done is considered Day 0. Therefore, if a test is done on a Monday, the Monday four weeks later would be considered Day 28. This allows for efficient patient scheduling without exceeding the guidelines. If Day 28 or 42 falls on a weekend or holiday, the limit may be extended to the next working day.
* All patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines.

Exclusion Criteria:

* Patients with the clinical diagnosis of congestive heart failure or angina pectoris are NOT eligible.
* Pregnant or nursing women may not participate due to the possibility of fetal harm or of harm to nursing infants from this treatment regimen. Women of reproductive potential may not participate unless they have agreed to use an effective contraceptive method. A urine pregnancy test is required for women of childbearing potential.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2005-10; Primary Completion 2013-09-04 (Actual); Study Completion 2013-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rita Mehta, M.D., Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (1):
- Chao Family Comprehensive Cancer Center, Orange, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at UCIMC by the following methods: referral for University of California Irvine Medical Center (UCIMC) inpatients or outpatients.
Groups:
- Chemotherapy With GM-CSF: Doxorubicin and Cyclophosphamide (AC) with Granulocyte-macrophage colony-stimulating factor (GM-CSF) (days 4-13) Followed by Weekly Carboplatin/Nab- Paclitaxel
Period: Overall Study
Arm/Group | Chemotherapy With GM-CSF
Started | 43
Completed | 41
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Chemotherapy With GM-CSF
Number analyzed (Participants) | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 36
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 43

OUTCOME MEASURES:

1. Primary Outcome: Overall Clinical Response to the Dose Dense Regimen
Description: Measure clinical response rates in patients with breast cancer more than 2 cm and/or lymph node positive breast cancer treated with 2- 4 cycles of biweekly doxorubicin, cyclophosphamide with GMCSF (day 4-13) followed by weekly carboplatin/nab-paclitaxel given for 3 weeks, followed by 1 week of rest, for a total of 9-12 doses. (Her-2 positive patients, in addition, will receive Trastuzumab weekly (12-16 doses) and Her-2 negative patients will receive Bevacizumab (6-8 doses) q 2 weeks).
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy With GM-CSF
Number analyzed (Participants) | 43
Participants | 43

ADVERSE EVENTS:
Arm/Group | Chemotherapy With GM-CSF
Serious Adverse Events (participants affected / at risk) | 4/43
Other Adverse Events (participants affected / at risk) | 0/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy With GM-CSF (N=43)
Neutropenic fever (Immune system disorders) | 3 (3)
Cardio Vascular Disease (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No